CLINICAL TRIAL: NCT07215780
Title: SORE Study: Sitz Baths After Urogynecologic Reconstruction
Acronym: SORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000040422
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Organ Prolapse; Postoperative Pain Management; Gynecologic Surgeries
Keywords: Pelvic organ prolapse surgical repair
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: The study population will consist of adult patients undergoing native tissue surgical repair of pelvic organ prolapse at a Yale-affiliated hospital.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sitz baths plus usual care (Experimental): Warm water sitz baths plus usual care. 7-day nightly regimen of warm water soaks without additives.
  Interventions: Device: Sitz Bath
- Usual care (No Intervention): Care as usual

INTERVENTIONS:
Device: Sitz Bath — Warm water sitz bath, 7 nights, 10 minutes each
  Arms: Sitz baths plus usual care

SUMMARY:
The purpose of this study is to evaluate the utility of postoperative sitz baths in patient pain perception and recovery following surgical repair of prolapse. The SORE Study is a prospective, randomized controlled trial that aims to compare postoperative pain intensity one week after native tissue repair of pelvic organ prolapse for patients undergoing a sitz bath regimen versus usual care. Findings from this study may contribute to more robust, multimodal postoperative pain management plans if proven efficacious or, alternatively, reduce plastic medical waste and simplify postoperative pain plans if found to be ineffective.

DETAILED DESCRIPTION:
The primary objective of the SORE study is to compare postoperative pain intensity one week after native tissue repair of pelvic organ prolapse for patients undergoing a sitz bath regimen versus usual care.

The secondary objectives of this study are to evaluate patient satisfaction with pain management after native tissue prolapse repair (and specifically posterior repair and/or perineorrhaphy), patient-reported opioid requirements, healthcare utilization, postoperative pain plan adherence, and incisional healing and complications between those undergoing a sitz bath regimen versus usual care.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years of age at time of surgery
* English or Spanish-speaking
* Documentation of pelvic organ prolapse as evidenced by Stage 2, 3, or 4 prolapse on preoperative Pelvic Organ Prolapse Quantification system (POP-Q) examination
* Surgery to be performed by a urogynecologist
* Ambulatory or inpatient surgery acceptable

Exclusion Criteria:

* Mesh-augmented prolapse repair (robotic, laparoscopic, or open sacrocolpopexy or sacrohysteropexy, vaginal mesh)
* Urogynecologic surgery without prolapse repair (i.e. midurethral sling, intravesicular botox, hysterectomy only)
* Suspected genital herpes simplex virus (HSV), molluscum contagiosum virus (MCV), condyloma acuminata, or vulvar/vaginal skin and soft tissue infection at recruitment by patient report
* Daily opioid use (short or long-acting)
* Concurrent non-urogynecologic surgery (i.e. rectopexy, staging or debulking for malignancy)
* Lack of access to operative report
* Pregnant (as determined by positive urine pregnancy test on the day of surgery via standard testing or current pregnancy documented in the preoperative note)
* Incarcerated
* Unable to give consent/conserved
* Unable to complete study intervention or assessment per investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Pain Intensity (PROMIS-PI) short form 3a questionnaire | Day 7 Post surgery
  Pain intensity will be assessed on a 15-point scale evaluating current, worst, and average pain on postoperative day 7 following prolapse repair and converted to a T- score using general population data. Higher scores indicate increased pain intensity.

SECONDARY OUTCOMES:
Mean score patient satisfaction | Day 7 Post surgery
  Satisfaction with postoperative pain management on a 0-100 mm visual analog scale
Mean Oxycodone use | Day 7 Post surgery
  Mean number of oxycodone tablets used postoperatively
Comfort with postoperative pain plan | Day 7 Post surgery
  Participant comfort level with managing postoperative multimodal pain plan on a 5-point Likert scale (1 = very uncomfortable, 5 = very comfortable)
Comfort with postoperative pain plan using Sitz bath | Day 7 Post surgery
  Participant comfort with sitz bath setup and cleanup, accessibility to bathroom use, physical comfort during and after use of sitz bath on a 5-point Likert scale (1 = very uncomfortable, 5 = very comfortable)
Sitz bath use- Adherence | Day 7 Post surgery
  Total use of sitz baths in minutes
Barriers to use- Adherence | Day 7 Post surgery
  Number of barriers to use perceived by self-report
Number of participants with rare adverse effects | Day 7 Post surgery
  Number of participants with any rare adverse effects per protocol
Mean Opioid use | Day 7 Post surgery
  Mean number of requests for opioid refills postoperatively
Mean number of calls regarding pain | Up to Day 90 Post surgery
  Mean number of calls or messages for postoperative pain within 90 days of surgery via review of medical record
Mean number of Emergency Department visits | Up to Day 90 Post surgery
  Mean number of emergency department visits within 90 days of surgery via review of medical record

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ringel, MD, MS, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Lawrence + Memorial Hospital, New London, Connecticut

IPD SHARING:
Plan to Share IPD: No